CLINICAL TRIAL: NCT03779035
Title: Adjuvant Chemotherapy With Gemcitabine and Capecitabine Compared to Capecitabine for Biliary Tract Cancer After Curative Resection
Brief Title: Adjuvant Chemotherapy for Biliary Tract Cancer After Curative Resection
Acronym: AdBTC-1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK2017144
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Cholangiocarcinoma; Gall Bladder Carcinoma
Keywords: adjuvant chemotherapy; cholangiocarcinoma; invasive gall bladder carcinoma; overall survival; disease free survival; Gemcitabine; Capecitabine
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms | interventions — Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gemcitabine plus Capecitabine (Experimental): Gemcitabine (1000 mg per square meter) on days 1 and 8 Capecitabine (1250 mg per square meter) twice a day on days 1-14. Treatment repeats every 3 weeks for 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine; Drug: Capecitabine
- Capecitabine (Active Comparator): Capecitabine (1250 mg per square meter) twice a day on days 1-14. Treatment repeats every 3 weeks for 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Gemcitabine — 1000mg/m2
  Arms: Gemcitabine plus Capecitabine
Drug: Capecitabine — 1250mg/m2

SUMMARY:
This prospective, open-Label, comparative, randomized, controlled phase III trial was designed to compare the clinical performance of gemcitabine with capecitabine vs. capecitabine alone for patients with biliary tract cancer (BTC) after curative resection.

DETAILED DESCRIPTION:
Currently, complete surgical resection represents the only potentially curative treatment option for cholangiocarcinoma (CCA, including intrahepatic, hilar and distal CCA) and gallbladder carcinoma (GBCA). Because of high rates of disease recurrence and poor survival rates following surgical resection, postoperative treatment have been considered to improve patient survival after resection of BTC. The systematic review showed a beneficial impact of adjuvant treatment in BTC, particularly in patients with involved lymph nodes or resection margins and distal or hilar CCA. However, in regard of the paucity of randomized data, current guidelines recommend inclusion in clinical trials.

Previously, the data of the BILCAP trial showed an improvement in median overall survival for capecitabine compared to observation alone for BTC, indicating capecitabine as the new standard postoperative treatment after curative resection of BTC.

Previous phase II studies for advanced BTC showed superiority of the combination gemcitabine/ capecitabine regimen vs. the capecitabine monotherapy, the median OS was 12.7-14 vs. 7.9 months.

Based on these data, this AdBTC trial will was designed to compare the clinical performance of gemcitabine with capecitabine vs. capecitabine alone for patients with biliary tract cancer (BTC) after curative resection, aiming for superiority of the combination regimen vs. the oral monotherapy. This will be based on the BILCAP protocol, applying the similar dosing, assessments and dose modifications.

The primary endpoint is DFS and secondary endpoints include recurrence free survival, OS, safety and tolerability of adjuvant CTx, quality of life, and patterns of disease recurrence.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed biliary tract cancer (including intrahepatic, extrahepatic, hilar cholangiocarcinoma or muscle invasive gallbladder cancer or cancer of the distal bile duct)
* Must have undergone a radical surgical approach which includes liver resection, pancreatic resection, or less commonly both
* Patients with pathological evidence of microscopic involvement of the margins of the excised specimen are eligible as long as resection is macroscopically complete
* Must be able to start treatment within 12 weeks of surgery
* No pancreatic or periampullary cancer
* No mucosal gallbladder cancer

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Urea < 1.5 times upper limit of normal (ULN)
* Creatinine < 1.5 times ULN
* Glomerular filtration rate ≥ 60 mL/min (if < 60 mL/min, adequate renal function for capecitabine must be confirmed by isotope EDTA)
* Hemoglobin ≥ 10 g/dL
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 3 times ULN
* ALT and AST ≤ 5 times ULN
* Adequate surgical biliary drainage with no evidence of infection
* Not pregnant or nursing
* Negative pregnancy test for women of childbearing age and childbearing potential
* Fertile patients must use effective contraception during study treatment and for at least 3 months after study treatment has ended
* Must provide written informed consent
* No history of other malignant diseases within the past 5 years
* No serious coexisting medical condition likely to interfere with protocol treatment, including a potential serious infection
* No evidence of significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial
* No psychological, familial, sociological, or geographical factors considered likely to preclude study compliance
* No other serious uncontrolled medical conditions
* No unresolved biliary tree obstruction

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Completely recovered from prior surgery
* No use of other investigational agents within 28 days prior to and during study treatment
* No prior chemotherapy or radiotherapy for biliary tract cancer
* No other concurrent anticancer chemotherapy, radiotherapy, or investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2018-12-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) rate | at 24 months
  DFS

SECONDARY OUTCOMES:
Overall survival (OS) rate | at 24 months
  OS
Disease free survival (DFS) rate | at 60 months
  DFS
Overall survival (OS) rate | at 60 months
  OS
The rate of patients with hepatic or locoregional recurrence | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Insititute and Hospital, Tianjin, Tianjin Municipality, China